CLINICAL TRIAL: NCT01319253
Title: Comparator Trial Evaluating Microbiological Resistance and Clinical Efficacy in Patients Using Alternation Therapy of Inhaled Antibiotics
Brief Title: A Comparator Study Evaluating Microbiological Resistance and Effects of Alternating Inhaled Antibiotic Therapies
Status: Completed | Type: Observational
Sponsor: Indiana University (Other)
Collaborators: Gilead Sciences (Industry)
Responsible Party: Principal Investigator, Michelle Howenstine, Professor of Clinical Pediatrics, Indiana University
Other Study IDs: HOWEN-ANDER-001
Record Dates: First submitted 2011-03-18; First posted 2011-03-21 (Estimated); Last update posted 2015-11-06 (Estimated); Status verified 2015-11

CONDITIONS: Cystic Fibrosis; Pseudomonas Aeruginosa
Keywords: Cystic Fibrosis; Pseudomonas aeruginosa
MeSH Terms: conditions — Cystic Fibrosis; Pseudomonas Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Cayston Only Cohort: This cohort will be on a previously established medication regiment of Cayston inhaled antibiotic alternating regimen every other month.
- Tobi Only Cohort: This Cohort will be on a previously established medication regiment that includes Tobi inhaled antibiotic regimen alternating every other month.
- Cayston and Tobi Cohort: This Cohort will be on a previously established medication regiment that includes Cayston and Tobi inhaled antibiotic alternating every other month

SUMMARY:
This is a pilot study of inhaled antibiotic regimens is a pilot study examining clinical and laboratory endpoints of patients on inhaled antibiotic treatments. We hypothesize that alternation therapy utilizing Cayston and Tobi will inhibit antibiotic resistance and that alternation therapy will result in a decreased incidence of antibiotic resistance to Cystic Fibrosis (CF) microbial isolates. The long term strategic goal is to develop a model biometric system for selecting a patient's optimal inhaled antibiotic regimen by utilizing clinical and microbiological parameters.

ELIGIBILITY:
Inclusion Criteria:

* > or = to 6 years of age
* Documentation of Cf diagnosis
* History of PA present in sputum, on a least one occasion, during the 12 months prior to Visit 1.
* Currently on inhaled antibiotic regiment
* Must be able to provide written informed consent or assent prior to any study related procedures
* Ability to expectorate sputum
* Ability ro perform reproducible pulmonary function test

Exclusion Criteria:

* Administration of any IV or oral antipseudomonal antibiotic within 28 days prior to Visit 1
* Any serious or active medical or psychiatric illness, which in the opinion of the investigator, woud interfere with participant treatment, assessment, or compliance with the protocol
* Current enrollment in an interventional clinical trial

Min Age: 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Primary care clinic
Sampling Method: Non-Probability Sample
Enrollment: 27 (Actual)
Dates: Start 2011-03; Primary Completion 2012-07 (Actual); Study Completion 2015-10 (Actual)

PRIMARY OUTCOMES:
Antibiotic Resistance Profiles | Every three months within a 12 month period
  The primary endpoint will be a change in the microbial resistance profile of pseudomonas aeruginosa (PA)isolates, change in PA sputum density, minimum inhibitory concentration of aztreonam and tobramycin for PA and the appearance or disappearance of other pathogens.

SECONDARY OUTCOMES:
Clinical Symptoms | Every 3 months within a 12 month period
  Secondary endpoint will be the change in clinical symptoms as assessed by the respiratory symptoms domain of the Cystic Fibrosis Questionnaire -Revised (CFQ-R),changes in pulmonary function Forced Exhaled Volume 1 second (FEV1) and change in frequency of hospitalizations or need for intravenous antibiotics.

CONTACTS AND LOCATIONS:
Overall Officials: Michelle S Howenstine, MD, Principal Investigator — Indiana University; Gregory Anderson, PhD, Principal Investigator — Indiana University
Locations (1):
- Indiana University, Indianapolis, Indiana, United States